CLINICAL TRIAL: NCT05505942
Title: Increasing Physical Activity Among Persons Living With HIV Engaged in Unhealthy Drinking
Brief Title: Physical Activity for PLWH and Unhealthy Drinking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-42543; 1P01AA029546-01 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HIV; Physical Inactivity; Unhealthy Alcohol Use
Keywords: Lifestyle physical activity (LPA); Fitbit; Telehealth; Unhealthy drinking; Ecological momentary assessment
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomization procedures to the two groups will apply sex at birth (male/female) and body mass index (greater than or equal to 30 or less than 30) as blocking variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Physical Activity (LPA) (Experimental): The LPA arm will receive 7 LPA sessions with a trained interventionist to assist in adding LPA to the participant's routine.
  Interventions: Behavioral: LPA Sessions
- Fitbit Only (Active Comparator): The Fitbit only arm will receive only brief check in phone calls and only related to assisting with any Fitbit functioning issues.
  Interventions: Other: Fitbit Only

INTERVENTIONS:
Behavioral: LPA Sessions — A study interventionist will conduct phone/video sessions and provide information regarding the acute and long-term psychological and physical benefits of increasing PA. Participants will be introduced to the concept of utilizing brief bouts of PA as a coping strategy for managing emotions and urges to drink alcohol "in-the-moment". Participants will also be given information on the public health guidelines for PA (and how these translate into step counts) as well as how to determine if their PA is moderate intensity (e.g., measuring heart rate and identifying rate of perceived exertion). Study clinicians will also orient participants to the proper use of the Fitbit activity tracker and tips for self-monitoring step counts with the tracker and on the app and/or website.
  Arms: Lifestyle Physical Activity (LPA)
Other: Fitbit Only — Interventionists will provide participants information about the proper use of the Fitbit activity tracker and offer tips for self-monitoring step counts with the tracker and on the app and/or website.
  Arms: Fitbit Only

SUMMARY:
Brief Summary: Alcohol use disorder (AUD) is a significant and costly public health problem that affects one-third of the U.S. population in their lifetime. Specifically, unhealthy alcohol use is common among persons living with HIV (PLWH) and increases the risk of developing negative outcomes. Antiretroviral therapy (ART) has shown increasing life expectancy and decreased HIV-related deaths, leading to a growing older adult HIV population. Yet, HIV accelerates the aging process and increases the risk for numerous chronic health conditions that compromise physical and mental health functioning and quality of life. Thus, PLWH continue to have shorter life expectancies relative to the general population and these multimorbidities explain this increased risk. In this context, unhealthy alcohol use among PLWH can further increase the risk for negative outcomes.

Physical activity (PA) interventions can be used as an effective way to address unhealthy alcohol use among PLWH. Previous PA interventions have shown low generalizability and high loss to follow-up. Therefore, an intervention that is home-based, including lifestyle physical activity (LPA) with mobile health-delivered components is designed following the physical activity (PA) paradigm.

Participants in this randomized controlled trial will be assigned to one of two study arms -- either the LPA or Fitbit Only intervention - both lasting 12-weeks. Both study arms will utilize a Fitbit to track daily step counts.

In addition to utilizing a Fitbit, the LPA arm will receive 7 LPA sessions with a trained interventionist to assist in adding LPA to the participant's routine.

The Fitbit only arm will receive only brief check-in phone calls and only related to assisting with any Fitbit functioning issues.

Follow-up assessments will take place at 3 and 6 months.

DETAILED DESCRIPTION:
Primary Aims - Physical Activity and Drinking Outcomes

To test the efficacy of a 12-week LPA intervention among low-active, PLWH engaged in unhealthy drinking. Participants will be randomly assigned to either: (a) LPA or (b) Fitbit Only control condition. Relative to Fitbit Only, the investigators hypothesize that:

1. LPA will demonstrate decreases in unhealthy drinking (i.e., drinks/week) end-of-treatment (EOT) and 3 months later (i.e., 6-month follow-up).
2. LPA will demonstrate higher objective-determined physical activity engagement (i.e., steps/day) at the EOT and at the 6-month follow-up.

Secondary Aims - Physical and Mental Health Functioning Outcomes Relative to Fitbit Only or LPA will result in decreased negative affect and sedentary behavior (i.e., minutes spent sitting/day), heavy drinking days, alcohol-related problems, and increases in adaptive coping, PA self-efficacy, PA motivation, and physical/mental functioning at EOT and 6-month follow-ups.

Tertiary Aims - Examining Mechanisms

1. Decreases in negative affect and increases in adaptive coping during the intervention period will mediate the relationship between LPA and drinking outcomes at the 6-month follow-up
2. Increases in PA self-efficacy and motivation will mediate the effect of LPA on PA engagement
3. Utilizing Ecological momentary assessment (EMA) and Fitbit data, we hypothesize higher negative affect and urges to drink earlier in the day is more likely to increase the likelihood of engaging in bouts of PA later in the day at EOT, relative to baseline, and among persons randomized to LPA versus Fitbit Only.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to confirm HIV diagnosis either through visual evidence of ART medication or medical record
* Engaged in unhealthy drinking, defined as: >7 drinks for women / > 14 drinks for men per week OR ≥ 3 drinks for women / ≥4 drinks for men on one occasion in the past month.
* Have a smartphone
* Considered low active: 150 minutes or less of average weekly physical activity
* Lives in the USA
* Has a U.S. mailing address

Exclusion Criteria:

* History of bipolar, schizophrenia, schizoaffective disorder or mania per self report.
* History of withdrawal-related seizures or delirium tremens per self report.
* Current non-pharmacological treatment for alcohol use disorder.
* Unable to provide one or more individuals for follow up contact.
* Current DSM-5 diagnosis of anorexia or bulimia nervosa per self report.
* Marked organic impairment according to responses to the diagnostic assessments
* Physical or medical problems that would not allow safe participation in a program of moderate intensity PA
* Individual who is unwilling to provide their sex at birth
* Limited or non-readers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in steps per day at 6-month follow up | 6 months
  Physical activity (PA) will be assessed via steps per day as collected by a participant's Fitbit.
Change in number of alcohol drinks consumed per week | 6 months
  Assessed by the Timeline Follow Back (TLFB-30) which is a is a calendar that allows an assessor to obtain an estimate of an individual's daily drinking habits over a 30-day time period.

SECONDARY OUTCOMES:
Change in steps per day at 3-month follow up | 3 months
  Physical activity (PA) will be assessed via steps per day as collected by a participant's Fitbit.
Change in alcohol drinks consumed per week | baseline
  Assessed by the Timeline Follow Back (TLBF-30) which is a is a calendar that allows a clinician to obtain an estimate of an individual's daily drinking habits over a given time period.
Changes in theoretically-relevant psychosocial factors including: negative affect, physical activity self-efficacy, physical activity motivation, alcohol-related problems, and time spent sitting | 3 months
  Assessed via self-report measures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Boston University, School of Public Health - Health Law Policy & Management; Lisa Quintiliani, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Boston University, Department of Medicine, remote research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No